CLINICAL TRIAL: NCT03674047
Title: A Phase II Study of Ruxolitinib for Bronchiolitis Obliterans Syndrome (BOS) After Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: Ruxolitinib for Bronchiolitis Obliterans Syndrome (BOS) After Allogeneic Hematopoietic Cell Transplantation (HCT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Zachariah Michael DeFilipp, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-265
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Other Cancer
Keywords: Hematopoietic Cell Transplantation
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- newly-diagnosed BOS (Experimental): -Participants will take ruxolitinib twice every day
  Interventions: Drug: ruxolitinib
- Established BOS (Experimental): -Participants will take ruxolitinib twice every day
  Interventions: Drug: ruxolitinib

INTERVENTIONS:
Drug: ruxolitinib — Ruxolitinib blocks certain proteins called tyrosine kinases. Specifically, it blocks tyrosine kinases called JAK2. it's believe that ruxolitinib may lower the rate of GVHD through its ability to block the JAK2 pathway since this pathway can lead to inflammation in the body
  Other Names: Jakafi

SUMMARY:
This research study is studying a drug as a possible treatment for Bronchiolitis Obliterans Syndrome (BOS) after having an Allogeneic Hematopoietic Cell Transplantation (HCT).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved ruxolitinib for this specific disease but it has been approved for other uses.

In this study the investigators are assessing the safety and effectiveness of ruxolitinib when given to participants who have been diagnosed with BOS after HCT. BOS is a sign/symptom of chronic Graft-vs-Host Disease (GVHD), a condition in which cells from the donor's tissue attack the organs after HCT occurs.

Ruxolitinib blocks certain proteins called tyrosine kinases. Specifically, it blocks tyrosine kinases called JAK2. The investigators believe that ruxolitinib may lower the rate of GVHD through its ability to block the JAK2 pathway since this pathway can lead to inflammation in the body.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BOS after HCT defined when all of the following criteria are met (as defined by the 2014 NIH criteria):

  * FEV1/VC < 0.7 or the 5th percentile of predicted.
  * FEV1 = Forced Expiratory Volume in 1 second.
  * VC = Vital Capacity (Forced Vital Capacity "FVC" or Slow Vital Capacity "SVC", whichever is greater)
  * The 5th percentile of predicted is the lower limit of the 90% confidence interval.
  * For elderly patients, use the lower limits of normal defined according to NHANESIII calculations.
  * FEV1 <75% of predicted with ≥ 10% absolute decline over less than 2 years. FEV1 should not correct to >75% of predicted with albuterol, and the absolute decline for the corrected values should still remain ≥ 10% over 2 years. The remote comparator would be an evaluation of PFTs done within 2 years of the PFTs assessment being evaluated to determine eligibility.
  * Absence of active infection in the respiratory tract, documented with investigations directed by clinical symptoms, such as chest radiographs or computed tomographic scans or microbiologic cultures (sinus aspiration, upper respiratory tract viral screen, sputum culture, bronchoalveolar lavage).
  * One of the two supporting features of BOS:
  * Evidence of air trapping by expiratory CT or small airway thickening or bronchiectasis by high-resolution chest CT OR
  * Evidence of air trapping by PFTs: RV (Residual Volume) > 120% of predicted or RV/TLC elevated outside the 90% confidence interval (RV/Total Lung Capacity).
* Life expectancy > 6 months at the time of enrollment as judged by the enrolling investigator.
* Male or female; 18-75 years old.
* ECOG Performance Status 0-2.
* At least 4 weeks since initiation of the most recent systemic therapy for cGVHD or BOS
* All females of childbearing potential must have a negative serum or urine pregnancy test < 7 days before study drug administration.
* The ability to understand and willingness to sign a written consent document

Exclusion Criteria:

* Recurrent malignancy or disease progression requiring anticancer therapy.
* Currently receiving or have previously received ruxolitinib for chronic GVHD therapy.
* Known history of allergy to ruxolitinib or its excipients.
* Pregnant females or nursing mothers.
* Hepatic dysfunction: transaminases (ALT, AST) > 5X ULN and/or total bilirubin > 3X ULN.
* Hematologic dysfunction: absolute neutrophil count <1000/μL, platelet cout <50K, and/or Hgb < 8 g/dL.
* Renal dysfunction: calculated creatinine clearance < 40 mL/min (Cockcroft-Gault formula)
* Receipt of any non-FDA approved study medication within the last 4 weeks (This does not apply to use of FDA-approved drugs for an off-label indication).
* Presence of an active uncontrolled infection. An active uncontrolled infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without signs or symptoms will not be interpreted as an active uncontrolled infection.
* Known human immunodeficiency virus infection.
* Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Subjects with previous positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
* Severe organ dysfunction unrelated to underlying GVHD, including: Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction).
* Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy.
* Clinically active asthma (variable and recurring symptoms of airflow obstruction and bronchial hyper-responsiveness), chronic obstructive pulmonary disease, interstitial lung disease, or cryptogenic organizing pneumonia or other causes of restrictive lung disease such as neuromuscular weakness or diaphragmatic paralysis.
* Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with the study requirements.
* Uncontrolled substance abuse or psychiatric disorder.
* Deemed (by the local PI or the PFT lab) unable to reliably perform pulmonary function tests.
* Active smoker of cigarettes or marijuana.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
absolute FEV1 increase | 3 Months
  The proportion of participants with a sustained, absolute FEV1 increase by ≥ 10% after 3 months of treatment with ruxolitinib (compared to baseline measure prior to study enrollment) among participants with newly diagnosed Bronchiolitis Obliterans Syndrome BOS.
treatment failure, comparing 3-month FEV1 to baseline FEV1 | 3 Months
  The proportion of participants who do not experience a sustained, absolute decrease in FEV1 by ≥ 10% after 3 months of treatment with ruxolitinib (compared to baseline measure prior to study enrollment) among participants with established Bronchiolitis Obliterans Syndrome BOS.

SECONDARY OUTCOMES:
Change scores for PFT measurements | 1 Year
  Change in pulmonary function test (PFT) measurements.
Improvements in chronic GVHD organ manifestations | 3 and 6 Months
  Improvements in chronic GVHD organ manifestations will be categorized according to the NIH chronic GVHD consensus criteria.
Overall survival | 2 Years
cGVHD progression-free survival | 2 Years
  cGVHD progression-free survival is defined as the time from registration to the earlier of progression of chronic GVHD or death due to any cause. Participants alive without cGVHD progression are censored at the date of last disease evaluation.
The incidence and types of serious adverse events | From the start of treatment until 30 days after the end of treatment, up to 13 months total
  Adverse events are graded according to Common Terminology Criteria for Adverse Events (CTCAE v4).
The total systemic corticosteroid dose longitudinally over time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zachariah DeFilipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - City of Hope Cancer Center, Duarte, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeFilipp Z, Kim HT, Cheng GS, Hamilton BK, Chhabra S, Hamadani M, Sandhu KS, Perez L, Lee CJ, Brennan TL, Garrelts C, Brown BM, Gallagher K, Newcomb RA, El-Jawahri A, Chen YB. A phase 2 multicenter trial of ruxolitinib to treat bronchiolitis obliterans syndrome after allogeneic HCT. Blood Adv. 2025 Jan 28;9(2):244-253. doi: 10.1182/bloodadvances.2024014000. PMID 39365992